CLINICAL TRIAL: NCT02881424
Title: Study of Familiarity in Alcohol Dependence : an Hyperfamiliarity for Faces
Brief Title: Study of Familiarity in Alcohol Dependence
Acronym: FALCO
Status: Terminated | Type: Observational
Sponsor: University Hospital, Lille (Other)
Responsible Party: Sponsor
Other Study IDs: 2014_51; 2014-A01761-46 (Other: ID-RCB number, ANSM)
Record Dates: First submitted 2016-08-17; First posted 2016-08-29 (Estimated); Last update posted 2018-10-15 (Actual); Status verified 2018-10

CONDITIONS: Alcohol Dependence
Keywords: Familiarity; Recollection; Face Recognition; Alcohol dependence; Social cognition
MeSH Terms: conditions — Alcoholism

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- alcohol-dependent patients: a group of 34 alcohol-dependent patients, currently abstinent
- healthy controls: a group of control subjects, without neurologic or psychiatric disease, matched for age and sex with the alcohol-dependent participants

SUMMARY:
Background:

Alcohol-dependence is a chronic disease with a high risk of relapse. The main therapeutic outcome relies on relapse prevention which seeks to identify high risk situations and individual's response to these situations especially the emotional response to social environment. Alcohol-dependence also induces cognitive impairments leading to social cognition impairments increasing the risk of relapse.

Familiarity is a key process in social interactions: it induces the feeling of prior knowledge of a stimulus without remembering consciously its identity. Followed by a second process based on the contribution of contextual information (recollection) familiarity allows face recognition.

Main aim:

Study of familiarity for faces in alcohol-dependence

Secondary objectives:

Highlighting correlations between familiarity impairments and clinical outcomes

DETAILED DESCRIPTION:
Familiarity will be tested by a specific familiarity task using an original paradigm. This paradigm allows the analysis of familiarity as a quantitative process as well as the analysis of personal familiarity to each subject. Three familiar and three unfamiliar faces are morphed in pairs for each participant. The displayed stimuli for each pair of faces are ten morphs with 5 to 95% of familiar face increasing by 10%. Participants are asked to press a button if the displayed stimulus seems familiar. At the end of the task each participant is asked to name the identity of the familiar faces (true or false recognitions, true or false omissions).

Each participant will undergo 2 visits.

* First visit:

  * Checking the inclusion and non-inclusion criteria
  * Clinical report and alcohol consumption evaluation
  * Standardized psychiatric interview (Mini International Neuropsychiatric Interview - MINI)
  * Neuropsychological tests (Montreal Cognitive Assessment - MoCA, "Batterie Rapide d'Efficience Frontale" - BREF, "Rappel Libre et Rappel Indicé à 16 items" - Grober & Buschke 's test - RL/RI 16)
* Second visit:

  * Checking the non-consumption of alcohol and other drugs (cannabis, amphetamine, cocaine, methamphetamine, ecstasy, opioid)
  * Task of familiarity with a controlling task
  * Social cognition test (Movie for the Assessment of Social Cognition - MASC)

ELIGIBILITY:
Inclusion Criteria:

* For all participants:

  * With normal vision with or without glasses
  * Understanding the Note of information and signing the consent form
* For alcohol-dependent patients:

  * Being diagnosed with severe alcohol addiction (according to DSM-5)
  * Currently abstinent
* For control subjects:

  * Exclusion of severe alcohol addiction's diagnosis (according to DSM-5)
  * Without antecedent or current neurologic disease
  * Without antecedent or current psychiatric disease
  * Non-taking psychotropic drugs

Exclusion Criteria:

* For all participants:

  * Pregnant or breast-feeding women
  * Cognitive impairment detected by a MoCA score inferior to < 26/30
  * Physically or mentally not able to pass the tests of the study
  * Taking an unauthorized drug the month before entering the study (other psychotropic drugs than the ones used for withdrawal or alcohol related complications for patients and any psychotropic drug for control subject)
  * Being diagnosed with a severe addiction other than to caffeine or tobacco (according to DSM-5)
  * Criteria for a plausible fetal alcohol syndrome
* For alcohol-dependent patients:

  * Being diagnosed with schizophrenia or bipolar disorder (according to DSM-5)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 34 participants will be included in 2 groups: one group of alcohol-dependent patients and another group of control subjects matched for age and sex.
Sampling Method: Non-Probability Sample
Enrollment: 42 (Actual)
Dates: Start 2015-03 (Actual); Primary Completion 2018-04 (Actual); Study Completion 2018-04 (Actual)

PRIMARY OUTCOMES:
Familiarity threshold | 3 years
  calculated from the psychometric function of each participant

SECONDARY OUTCOMES:
Alcohol consumption | 3 years
  alcohol consumption evaluation
MocA score | 3 years
  Score at the Montreal Cognitive Assessment
BREF score | 3 years
  neuropsychological score
RL/RI score | 3 years
  neuropsychological score
non-consumption of alcohol duration | 3 years
  non-consumption of alcohol duration
social cognition test | 3 years
  social cognition test score
concomitant treatment | 3 years
  concomitant treatment posology

CONTACTS AND LOCATIONS:
Overall Officials: Olivier COTTENCIN, MD, PhD, Principal Investigator — University Hospital, Lille
Locations (2):
- France (2):
  - University Hospital, Lille - CSAPA, Lille
  - University Hospital, Lille - Fontan 2, Lille

IPD SHARING:
Plan to Share IPD: No